CLINICAL TRIAL: NCT06987929
Title: A Randomised Controlled Trial Comparing the Efficacy of Ultrasound-guided Hydrodilatation With Intra-articular Corticosteroid Injection in the Treatment of Adhesive Capsulitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/2474
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Adhesive Capsulitis, Shoulder
Keywords: Adhesive capsulitis, corticosteroid, hydrodilatation, interventional studies, intra-articular agents, pain assessment and management, ultrasonography
MeSH Terms: conditions — Bursitis | interventions — Steroids

STUDY DESIGN:
Intervention Model Description: single-centre, prospective, open-label randomised controlled study (RCT)
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (Other)
  Interventions: Procedure: Intra-articular steroid injection (IAI)
- Hydrodilation (Active Comparator)
  Interventions: Procedure: Hydrodilatation injection

INTERVENTIONS:
Procedure: Hydrodilatation injection — During the procedure, the patient lie supine on an examination couch, with the affected arm in the modified Crass position. All injections were done under image guidance using a Philips EPIQ ultrasound machine with an L18-12 MHz linear array transducer, performed consecutively by 2 rheumatologists or 1 pain medicine anaesthetist, all trained in MSK US. Aseptic technique was used. The transducer was placed at the short axis of the supraspinatus tendon, and the rotator cuff interval and coracohumeral ligament (CHL) were identified. Local anaesthetic (1% lignocaine) was injected subcutaneously to the skin. The therapeutic medication consisted of a mixture of 40 mg triamcinolone (10 mg/ml concentration) and 5ml 1% lignocaine, which was diluted with sterile normal saline into a total of 20mls suspension. The injection was administered using a 22-G 2-inch needle (Stimuplex A) introduced below the CHL adjacent to the long head of biceps tendon, in the in-plane view under US guidance.
  Arms: Hydrodilation
Procedure: Intra-articular steroid injection (IAI) — Intra-articular corticosteroid injection was performed as a control group. The posterior shoulder approach was used. The patient was positioned in the lateral decubitus or semi-prone position with the affected shoulder at the uppermost position, elbow semi-flexed and the ipsilateral arm resting on a pillow for comfort and stability. The ultrasound transducer is positioned over the long axis of the myotendinous junction of the infraspinatous tendon to view the contours of the posterior glenoid labrum and posterior portion of the humeral head. The injectate was administered using a 21-G hypodermic needle. 40 mg triamcinolone (10 mg/ml concentration) mixed with 1ml of 1% lignocaine was injected into the posterior glenohumeral joint, under ultrasound-guidance. Any adverse reaction that occurred during the procedure was recorded. Following the procedure, the patient was advised to avoid overuse of the injected joint for 24 hours as part of post-injection care.
  Arms: Conventional Group

SUMMARY:
This study aims to evaluate the effectiveness of HD compared with intra-articular corticosteroid injection (IAI) in patients with adhesive capsulitis, with pain and function as the primary outcomes. We conducted a prospective, randomised controlled trial conducted in the Rheumatology department of a tertiary centre. Twenty patients with adhesive capsulitis were recruited and randomised equally to receive HD (n = 10), and IAI (n = 10). The primary outcome measures include Shoulder Pain and Disability Index (SPADI), QuickDASH questionnaire score, pain visual analogue scale (VAS) score, and range of motion (ROM) at 6-weeks post-intervention.

DETAILED DESCRIPTION:
Adhesive capsulits is a common shoulder condition that causes significant pain and loss of joint mobility, thus affecting the quality of life. If left untreated, the symptoms can impair the person's function and persist for a longer duration. Both hydrodilatation and standard steroid injection into the glenohumeral joint are well recognised forms of treatment, but there is no consensus on the best treatment approach for adhesive capsulitis. Hydrodilatation involves injecting a larger volume of solution (with steroid and local anaesthetic mixed), into the space within the rotator cuff interval, leading to intra-articular distension of the joint capsule. The local anaesthetic used in the procedure provides immediate pain relief, while the long-term benefit comes from the resolution of the capsular stiffness and inflammation. This process stretches the capsule, resulting in adhesion breakdown and promoting the remodeling of the shoulder capsule, hence improving shoulder range of motion (ROM), especially in those with limited mobility due to the capsular tightening. This study aims to evaluate the effectiveness of HD compared with intra-articular corticosteroid injection (IAI) in patients with adhesive capsulitis, with pain and function as the primary outcomes. We conducted a prospective, randomised controlled trial conducted in the Rheumatology department of a tertiary centre. Twenty patients with adhesive capsulitis were recruited and randomised equally to receive HD (n = 10), and IAI (n = 10). The primary outcome measures include Shoulder Pain and Disability Index (SPADI), QuickDASH questionnaire score, pain visual analogue scale (VAS) score, and range of motion (ROM) at 6-weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. adhesive capsulitis or frozen shoulder, diagnosed clinically, with or without imaging,
2. persistent symptoms of pain and restricted ROM for at least 3 months, despite conservative management with physiotherapy and/or analgesia

Exclusion Criteria:

1. previous surgery or shoulder implants of the affected shoulder,
2. history of recent trauma or fracture involving the affected shoulder,
3. age below 21 years,
4. pregnant women,
5. any evidence of ongoing active systemic inflammatory arthritis,
6. allergy to any of the injectates,
7. patients on anticoagulation (warfarin or direct oral anticoagulant),
8. received any joint injection in the past 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 6 weeks
  SPADI: self-reported questionnaire by patient on pain and disability.
QuickDASH score | 6 weeks
  self-reported questionnaire by patient on upper extremity disability
Pain score | 6 weeks
  self-reported by patient using visual analogue scale (VAS).
Active and passive range of motions (ROM): | 6 weeks
  measured by investigators blinded to the treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Chew Li Ching, Principal Investigator — Singapore General Hospital
Locations (1):
- Autoimmunity and Rheumatology Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The authors adhered to the consort recommendations for clinical trials. Study Protocol may be shared with other researchers by authors upon request.